CLINICAL TRIAL: NCT07400211
Title: Non-invasive Molecular Diagnostics for Inflammatory Bowel Disease : A Genetic and Biomarkers Study
Brief Title: Diagnosis of Inflammatory Bowel Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sandy Sameh Naguib Fanous, Doctor, Assiut University
Other Study IDs: Non-invasive diagnosis of IBD
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Inflammatory Bowel Disease (IBD)
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with inflammatory bowel disease
- Healthy normal persons

SUMMARY:
* To quantify the expression of Nuclear enriched abundant transcript 1 (NEAT1) and Anti-sense Non RNA in the INLK4 locus (ANRIL) to determine their potential role as non invasive diagnostic biomarkers in inflammatory bowel disease.
* To evaluate the correlation between the studied biomarkers and both the clinical presentation of the patients and the inflammatory mediators like Nuclear factor κB (NF-KB) signaling pathway.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic inflammatory disorder affecting the gastrointestinal tract and is characterized by a progressive and unpredictable disease course. There has been a global rise in the incidence of IBD over the last few decades. Considering the chronic, progressive nature of IBD and the costliness of its treatment, the rise of IBD entails a growing socioeconomic burden. A growing body of evidence suggests that IBD may be the result of an interaction between genetic factors, environmental factors, life style factors as diet, antibiotics, intestinal barrier dysfunctions and altered microbes.

According to a large meta-analysis of population-based studies (2000-2022) The global prevalence rates of IBD was 229.7 per 100,000 persons and the incidence was 9.7 per 100,000 persons. Europe had the highest prevalence rates of IBD while the highest IBD incidence was seen in Oceania. Research in the Arab world suggests that the IBD prevalence in Arab countries increased from ~28.9 to ~34 cases per 100,000 between 2009 and 2019, with Egypt as one of the leading countries producing IBD research output. According to a recent global burden study (1990-2021), the absolute number of deaths attributed to IBD nearly doubled: from ~21,418 in 1990 to ~42,422 in 2021 - reflecting growing numbers of people living with IBD.

It is characterized by remission and exacerbation course. Bloody stools, abdominal pain, weight loss, chronic diarrhea, and the presence of immune-mediated extra-intestinal manifestations represent the disease's symptoms.

Over time, severe inflammation within the intestine can lead to serious complications, including ulcers, narrowing of the intestinal lumen, and even perforations. Notably, IBD can cause considerable damage to the digestive system, resulting in substantial tissue injury, reduced intestinal functionality, associated disability, and a state of systemic inflammation that may impact the individual's overall health. Also, Patients with inflammatory bowel disease have an increased risk of developing colorectal cancer.

Inflammatory bowel disease manifests primarily in two major forms: Crohn's disease (CD) and ulcerative colitis (UC) . Crohn's disease typically exhibits lesions in the ileum and colon, characterized by intermittent inflammatory changes of the permeable wall while Ulcerative colitis predominately develops on the mucosal surface of the rectum, displaying continuous inflammatory foci.

The causative genes responsible for IBD remain incompletely characterized, highlighting the necessity for a thorough investigation of crucial molecular signatures involved in its development, which may provide potential avenues for effective therapies. In recent years, there has been a significant expansion in the era of RNA biology, showing the sophisticated mechanisms of gene regulation that extend far beyond the conventional protein-coding genes. While messenger RNAs (mRNAs) are transcribed and translated into proteins, most of the genome is transcribed into RNA molecules known as non-coding RNAs (ncRNAs) that do not ultimately translate into proteins.

Over 70% of genetic associations in IBD occur in the noncoding regions of the genome. The major classes of ncRNAs that have gained increased research attention are long non-coding RNAs (lncRNAs), microRNAs (miRNAs), and circular RNAs (circRNAs). Long noncoding RNA are noncoding RNAs (not get translated into protein) with a length of more than 200 base pairs , and contribute to the etiology of various diseases such as respiratory diseases, inflammatory diseases and tumors. lncRNAs are major players in the inflammatory pathway as they have crucial roles in not only expression but also differentiation of cytokines and immune cells, respectively.

Nuclear enriched abundant transcript 1 (NEAT1) is long noncoding RNA that is a key component in building the ribo-riboprotein complex to regulate DNA-mediated activation of innate immune responses and has also been found to play an important role in innate immune responses. It targets numerous genomic regions in various cells, mainly involving active genes, revealing that it is a regulator for plenty of active genes and signal pathways. It is involved in the development of colitis by acting on miR-204-5p axis through activating PI3K-AKT signaling pathway and the NF-κB signaling pathway leading to increase of Interleukin-6 (IL-6) , Imterleukin-1B (IL-1B) and Tumor necrosis factor-a (TNF-a) that result in inflammation and cell apoptosis .

Anti-sense Non RNA in the INLK4 locus (ANRIL) is long non coding RNA that doesn't encode a protein; instead, it regulates gene expression at transcriptional, epigenetic, and post-transcriptional levels . It has a pro-inflammatory role in many inflammatory and immune diseases as Coronary artery disease, Chronic kidney disease and Inflammatory bowel disease. In IBD, it mediates nuclear factor κB (NF-κB) to influence inflammation through its effects on intestinal epithelial cells, besides providing future clues for clinical diagnosis. It activates NF-ΚB leading to increase of IL-6 , IL-1B and TNF-a that result in cell apoptosis . Also, Up-regulation of ANRIL could decrease the expression of miR-199a and increase the number of apoptotic cells.

Nuclear factor kappa B (NF-KB) expression is accompanied by increased production of pro-inﬂammatory cytokines, such as TNF-α, IL-1 and IL-6, due to the actions of NF-kB in expanding the capacity of these cells to produce inﬂammatory mediators. Predominantly, the NF-kB derived pro-inﬂammatory cytokines are responsible for two mechanisms involved in the development of IBD lesions. Firstly, the produced pro-inﬂammatory cytokines directly mediate mucosal tissue damage by principally up-regulation of matrix metalloproteinases production and secretion in the intestinal lumen. Secondly, NF-kB derived pro-inﬂammatory cytokines also mediate the stimulation, activation, and differentiation of immunological cells derived from lamina propria of the bowel mucosa, resulting in chronic inﬂammation and, therefore, in the perpetuation of mucosal damage.

So the investigators will measure NEAT1 and ANRIL as diagnostic biomarkers for IBD together with the Inflammatory mediator NF-KB. This can be done by non invasive blood sample instead of the invasive endoscopic biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Newly histopathologicaly diagnosed IBD

Exclusion Criteria:

* Patients with serious complications as intestinal obstruction, perforation, polyps or colorectal carcinoma
* Patients who are taking NSAIDs or Immunosuppressive drugs
* Patients who are having other autoimmune disorders
* Patients with Chronic infections as TB or other diseases
* Patients with a history of allergy
* Pregnant or Lactating women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with inflammatory bowel disease
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
To quantify the expression of NEAT1 and ANRIL to determine their potential role as non invasive diagnostic biomarkers in inflammatory bowel disease. | Baseline
  Measure level of NEAT1 and ANRIL genes in blood samples of inflammatory bowel disease patients

SECONDARY OUTCOMES:
To evaluate the correlation between the studied biomarkers among the studied groups explored and both their clinical presentations and the inflammatory mediators like NF-KB signaling pathway. | Baseline
  To find the relation between the studied biomarkers (NEAT1 and ANRIL) and the inflammatory mediators like NF-KB signaling pathway.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laurindo LF, Santos AROD, Carvalho ACA, Bechara MD, Guiguer EL, Goulart RA, Vargas Sinatora R, Araujo AC, Barbalho SM. Phytochemicals and Regulation of NF-kB in Inflammatory Bowel Diseases: An Overview of In Vitro and In Vivo Effects. Metabolites. 2023 Jan 7;13(1):96. doi: 10.3390/metabo13010096. PMID 36677021
- [Background] Pan Y, Wang T, Zhao Z, Wei W, Yang X, Wang X, Xin W. Novel Insights into the Emerging Role of Neat1 and Its Effects Downstream in the Regulation of Inflammation. J Inflamm Res. 2022 Jan 26;15:557-571. doi: 10.2147/JIR.S338162. eCollection 2022. PMID 35115805
- [Background] Walther K, Schulte LN. The role of lncRNAs in innate immunity and inflammation. RNA Biol. 2021 May;18(5):587-603. doi: 10.1080/15476286.2020.1845505. Epub 2020 Nov 19. PMID 33138685
- [Background] Mineo M, Lyons SM, Zdioruk M, von Spreckelsen N, Ferrer-Luna R, Ito H, Alayo QA, Kharel P, Giantini Larsen A, Fan WY, Auduong S, Grauwet K, Passaro C, Khalsa JK, Shah K, Reardon DA, Ligon KL, Beroukhim R, Nakashima H, Ivanov P, Anderson PJ, Lawler SE, Chiocca EA. Tumor Interferon Signaling Is Regulated by a lncRNA INCR1 Transcribed from the PD-L1 Locus. Mol Cell. 2020 Jun 18;78(6):1207-1223.e8. doi: 10.1016/j.molcel.2020.05.015. Epub 2020 Jun 5. PMID 32504554
- [Background] Leitao AL, Enguita FJ. A Structural View of miRNA Biogenesis and Function. Noncoding RNA. 2022 Jan 18;8(1):10. doi: 10.3390/ncrna8010010. PMID 35202084
- [Background] Johnson JL, Sargsyan D, Neiman EM, Hart A, Stojmirovic A, Kosoy R, Irizar H, Suarez-Farinas M, Song WM, Argmann C, Avey S, Shmuel-Galia L, Vierbuchen T, Bongers G, Sun Y, Edelstein L, Perrigoue J, Towne JE, Hall AO, Fitzgerald KA, Hoebe K. Gene coexpression networks reveal a broad role for lncRNAs in inflammatory bowel disease. JCI Insight. 2024 Feb 8;9(3):e168988. doi: 10.1172/jci.insight.168988. PMID 38329124
- [Background] Hossam Abdelmonem B, Kamal LT, Wardy LW, Ragheb M, Hanna MM, Elsharkawy M, Abdelnaser A. Non-coding RNAs: emerging biomarkers and therapeutic targets in cancer and inflammatory diseases. Front Oncol. 2025 Mar 10;15:1534862. doi: 10.3389/fonc.2025.1534862. eCollection 2025. PMID 40129920
- [Background] Luo Q, Wang J, Ge W, Li Z, Mao Y, Wang C, Zhang L. Exploration of the potential causative genes for inflammatory bowel disease: Transcriptome-wide association analysis, Mendelian randomization analysis and Bayesian colocalisation. Heliyon. 2024 Apr 6;10(7):e28944. doi: 10.1016/j.heliyon.2024.e28944. eCollection 2024 Apr 15. PMID 38617957
- [Background] Sato Y, Tsujinaka S, Miura T, Kitamura Y, Suzuki H, Shibata C. Inflammatory Bowel Disease and Colorectal Cancer: Epidemiology, Etiology, Surveillance, and Management. Cancers (Basel). 2023 Aug 17;15(16):4154. doi: 10.3390/cancers15164154. PMID 37627182
- [Background] Li T, Jing H, Gao X, Zhang T, Yao H, Zhang X, Zhang M. Identification of key genes as diagnostic biomarkers for IBD using bioinformatics and machine learning. J Transl Med. 2025 Jul 3;23(1):738. doi: 10.1186/s12967-025-06531-1. PMID 40611294
- [Background] Erfan R, Shaker OG, Khalil MAF, Mahmoud FAM, Gomaa MS, Abu-El-Azayem AK, Zaki OM, Ahmed AM, Samy A, Mohammed A. Circulating miR-199a and long noncoding-RNA ANRIL as Promising Diagnostic Biomarkers for Inflammatory Bowel Disease. Inflamm Bowel Dis. 2024 Sep 3;30(9):1500-1509. doi: 10.1093/ibd/izad210. PMID 38190238
- [Background] Lin D, Jin Y, Shao X, Xu Y, Ma G, Jiang Y, Xu Y, Jiang Y, Hu D. Global, regional, and national burden of inflammatory bowel disease, 1990-2021: Insights from the global burden of disease 2021. Int J Colorectal Dis. 2024 Sep 7;39(1):139. doi: 10.1007/s00384-024-04711-x. PMID 39243331
- [Background] AlMuhaidib S, Bzeizi K, AlAmeel T, Mosli M, Khoja B, Barakeh D, Alomaim WS, Alqahtani SA, Al-Bawardy B. A bibliometric analysis of inflammatory bowel disease research in the Arab world. Saudi J Gastroenterol. 2025 May 1;31(3):146-156. doi: 10.4103/sjg.sjg_303_24. Epub 2024 Dec 11. PMID 39660608
- [Background] Heydari K, Rahnavard M, Ghahramani S, Hoseini A, Alizadeh-Navaei R, Rafati S, Raei M, Vahidipour M, Salehi F, Motafeghi F, Neshat S, Moosazadeh M, Yousefi M, Pourali A, Rasouli K, Shokrirad S, Lotfi P, Beladi SA, Hadizadeh Neisanghalb M, Sheydaee F, Moghadam S. Global prevalence and incidence of inflammatory bowel disease: a systematic review and meta-analysis of population-based studies. Gastroenterol Hepatol Bed Bench. 2025;18(2):132-146. doi: 10.22037/ghfbb.v18i2.3105. PMID 40936779
- [Background] Hu Y, Lu Y, Fang Y, Zhang Q, Zheng Z, Zheng X, Ye X, Chen Y, Ding J, Yang J. Role of long non-coding RNA in inflammatory bowel disease. Front Immunol. 2024 Jun 4;15:1406538. doi: 10.3389/fimmu.2024.1406538. eCollection 2024. PMID 38895124
- [Background] Mak WY, Zhao M, Ng SC, Burisch J. The epidemiology of inflammatory bowel disease: East meets west. J Gastroenterol Hepatol. 2020 Mar;35(3):380-389. doi: 10.1111/jgh.14872. Epub 2019 Nov 24. PMID 31596960